CLINICAL TRIAL: NCT03175692
Title: Rapid Genetic Diagnosis Employing Next Generation Sequencing for Critical Illness in Infants and Children
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 201703073RINB
Record Dates: First submitted 2017-05-23; First posted 2017-06-05 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-05

CONDITIONS: Congenital Metabolic Disorder; Acute Disease
MeSH Terms: conditions — Metabolism, Inborn Errors; Acute Disease | interventions — Exome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Use blood or DBS to extract DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- critical illness in infants and children: Those infants and children who has congenital metabolism disorder or acute disorder.
  Interventions: Diagnostic Test: Whole Exome Sequencing

INTERVENTIONS:
Diagnostic Test: Whole Exome Sequencing — Using next generation sequencing to analysis patient's whole exome. To explore the pathogenic gene variation.

SUMMARY:
Under the joint efforts of genetic and intensive expert, to establish the high-throughput whole exon sequencing(WES) and analysis all the possible pathogenic genes. To provide patient with the appropriate treatment for genetic disease. Besides, it can identify the genetic factor of idiosyncrasy or susceptibility to explain the medical difficulties and give patients personalized advice.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients admitted to intensive care unit
* Infants with abnormal newborn screening result that is medical emergency

Exclusion Criteria:

* Participants or parents who cannot comply with study

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and newborn patients at National Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-06-14 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of whole exome sequencing in detecting causative mutations | 10 weeks

SECONDARY OUTCOMES:
Time frame of mutation identified after receipt of the sample | 10 weeks
Percentage of mutation identified within 7 days after receipt of the sample | 10 weeks
Changes in healthcare decision after disclosure of the result | 6 months
Parents/family's attitude about exome sequencing | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wuh-Liang Hwu, Principal Investigator — Department of Pediatrics and Medical Genetics, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No